CLINICAL TRIAL: NCT00755573
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Clinical and Experimental Pilot Study of Pregabalin in Patients With Chronic Pancreatitis
Brief Title: Pain and Chronic Pancreatitis - Clinical End Experimental Studies
Acronym: CPP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Asbjørn Drewes Professor, Department of Gastroenterology, Aalborg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081172/8967
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Pancreatitis
Keywords: Pain; Neuropathic pain
MeSH Terms: conditions — Pancreatitis, Chronic; Pain; Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator): Pregabalin 300 mg - 600 mg BID
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 300 mg - 600 mg BID
  Other Names: Lyrica
  Arms: Pregabalin
Drug: placebo — Regime as described for pregabalin
  Other Names: Inactive comparator (placebo)
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the effect of pregabalin in pain resulting from chronic pancreatitis. The effect will be investigated by means of questionnaires concerning the daily experience of pain and the general quality of life. Furthermore the patients will be invited to participate in experimental testing with a multimodal pain model. The experimental testing will include stimulation of the skin, muscle and visceral tissue. The results from the experimental part of the study may help us to understand the mechanisms of action of pregabalin in this patient population.

DETAILED DESCRIPTION:
Background and Rationale

The aetiology of pain in chronic pancreatitis remains to be elucidated. Therefore no common guidelines for the management of the pain exist and it is a topic of great discussion. The area is further complicated by the fact that only a few clinical trials have been carried out (Wilder-Smith et al. 1999). The best attempt to establish clear guidelines for the treatment of chronic pancreatitis is "American Gastroenterological Association Medical Position Statement: Treatment of Pain in Chronic Pancreatitis" (Warshaw et al. 1998). Initial treatment consists of low fat diet and non-narcotic analgesics, which can be supplemented by oral pancreatic enzymes and proton pump inhibitors. If an acceptable level of pain relief is not obtained with these drugs, only opioids remain for the management of pain. Opioids have a number of well-known adverse effects including elevation of smooth muscle tone (affecting gastrointestinal motility), toxicity in the central nervous system and especially induction of addiction. Many patients suffering from chronic pancreatitis have a history of alcoholic abuse making opioids, with their associated abuse potential, less suitable for these patients. Alternatives to medical treatment exist in the form of nerve blockade, lithotripsy and surgical treatment. However, results from studies of non-medical treatment modalities are equivocal and medical analgesic therapy must still be considered as the first choice in the management of painful chronic pancreatitis. Thus the importance of identifying potential new treatment regimes for the treatment of pain in chronic pancreatitis is clear.

In patients with chronic pancreatitis the pancreatic nerves have been found to have a greater diameter and the area innervated by a single nerve is smaller (Bockman et al. 1988). A neural genesis of pain therefore seems likely. The basis of the neurogenic generation of pain may be due to an altered expression of neuropeptides like SP and CGRP. The concentration of nerve growth factor (NGF) and its receptor TrkA is increased in inflammatory areas which may lead to an enhanced transcription of SP and CGRP, both of which are transmitters in the pain system (Di Sebatiano et al. 2003). Interestingly, the release of SP is known to be reduced by agents such as pregabalin.

Support for a neuropathic component of the pain of chronic pancreatitis is also found in clinical observations, where the pain is typically described as largely constant background pain with shooting, burning and lancinating episodes that may mimic that seen in peripheral neuropathies. Finally, evidence for central neuroplastic findings and strong descending inhibition, which may reflect the pain mechanisms in neuropathic pain have been found in recent studies (Dimcevski et al. 2006 and 2007). Thus inflammatory and "true" visceral pain components appear to play a role in pancreatic pain. Hence the potential to extrapolate from clinical trials demonstrating the activity of pregabalin in the treatment of neuropathic pain to the treatment of the possible neuropathic component of chronic pancreatitis is of great interest.

Central sensitization is an essential factor in the development of neuropathic pain (Baron 2001, Johnson et al. 2001) and in animal experiments the NMDA receptor has been shown to be involved in this process. Calcium plays a central role, as an increased influx of calcium into the neuron is observed when the NMDA receptor is activated. The enhanced concentration of intracellular calcium functions as a second messenger for a number of neurotransmitters and calcium thus contributes to the maintenance of the central sensitization (Nicholson 2000).

Pregabalin exerts a range of effects in pain transmission and although the precise mechanism of action is not completely understood, it likely involves the binding of the drug to calcium channels in the central nervous system (Ben-Menachem 2004). In animal experiments it has been shown that pregabalin primarily exerts its effect in the dorsal horn, where a reduced pain signal is seen. Pregabalin is a ligand of the α2-δ subunit of the voltage-gated calcium channel and binding of pregabalin to this site results in reduced calcium influx at the nerve terminals and therefore a reduced release of several excitatory neurotransmitters, including glutamate, substance P (SP), calcitonin-gene related peptide (CGRP) and noradrenaline. This may result in inhibition or reduction of the sensitization mentioned above. Moreover, this may be the basis for the analgesic effect. It has been shown, in animal experiments, that binding of pregabalin to calcium channels is able to counteract central sensitization in the dorsal horn.

The evidence for the clinical effect of pregabalin in neuropathic pain is substantial and is documented in a number of randomized clinical trials (Dworkin et al. 2003, Sabatowski et al. 2004, Rosenstock et al. 2004). The recommended dose for treating neuropatic pain is between 150 mg to 600 mg daily, which is similar to the dose chosen for this study. By the opinion of the principal investigator no clinically relevant medical interactions are described for pregabalin when administered for chronic pancratitis patients.

Pregabalin is absorbed in the small intestine by a saturable transporter (Piyapolrungroj et al. 2001). It is well known that pancreatitis patients suffer from malabsorption of fat and therefore frequently suffer from diarrhea. This could lead to changes in the mucosal surface in the small intestine, and possibly change the absorption of pregabalin. Drug absorption has never been investigated in patients suffering from pancreatitis and the simple and linear kinetics of pregabalin makes it possible to study how drug absorption may vary in these patients. A poorer absorption of drugs could partly explain why pain from pancreatitis is difficult to relieve.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18 and 75 years with a diagnosis of chronic pancreatitis diagnosed using the Mayo Clinic Diagnostic criteria criteria ((Layer P, Gastroenterology 1994;107:1481-1487]). Both diabetic and non-diabetic patients will be allowed to enter the study.
2. The patients must suffer from chronic abdominal pain typical for pancreatitis, meet the criteria for chronic pain (pain ≥ 3 days per week in at least 3 months) and must consider their pain as severe enough for medical treatment.
3. Personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.
4. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other trial procedures.

Exclusion Criteria:

1. Patients with evidence or history of medical or surgical disease of importance for this study as judged by investigator
2. Presence or history of major depression
3. Patients with previously diagnosed moderate to severe renal impairment. Patients with creatinine values > 2x ULN and/or with a significant change to their normal values should be excluded.
4. Patients with a screening 12-lead ECG demonstrating any of the following: heart rate >100 bpm, QRS duration >120 msec, QTc interval >450 msec, PR interval >210 msec, any clinically significant rhythm abnormality, any evidence of myocardial ischemia or injury.
5. Patients with any clinically significant laboratory abnormalities that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
6. Patients treated with pregabalin (Lyrica®) during the previous 4 months.
7. Treatment with an investigational drug within 4 months preceding the first dose of study medication of importance for this study as judged by investigator.
8. Female patients who are pregnant or lactating, or intend to become pregnant. Male patients who intend to father a child during the course of the study. A pregnancy test will be conducted at visit 1 and 3 to ensure that female patients are not pregnant during the study period. The investigator will have to ensure that fertile female patients use a safe contraception method during the study and for at least 35 hours after termination of the study period. The following methods are considered as safe contraception methods:

   * The pill
   * IUD
   * Gestagen Injection
   * Subdermal Implantation (Implanon)
   * Hormone vaginal ring
   * Transdermal Plaster
9. Patients unwilling or unable to comply with the lifestyle guidelines.
10. Patients must not suffer from generalized painful conditions other than chronic pancreatitis; however patients with localized painful disorders will be allowed to enter the study
11. Clinical significant illness within two weeks of participating in this study.
12. Involved in planning or conducting the study.
13. Hypersensitivity to pregabalin or any of its components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Patient pain diary based on the VAS score and different questionaries | Pain diary treatmentday -7 to +21. Questionaries are adressed 7 days prior to study medication and on day 21 during the study medication period
  The primary efficacy parameter to be evaluated is pain relief assessed using a patient pain diary based on the visual analog scale (VAS). Furthermore different questionnaires, including the modified brief pain inventory-short form (mBPI-sf), the painDETECT questionnaire (PD-Q) and patient global impression of change (PGIC)will be used to explore further aspects of pain character and influence on cognitive and affective components.

SECONDARY OUTCOMES:
Questionary addressing quality of life | Questionaries are adressed 7 days prior to study medication and on day 21 during the study medication period
  Secondary efficacy parameters are changes in quality of life compared to baseline level. The European Organization for research and treatment of cancer quality of life questionnaire (EORTC QOL-C30).Also the tolerability of the drug in this patient population will be compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, MD, PhD, Principal Investigator — Dapartment og Gastroenterology, Aalborg Hospital
Locations (2):
- Department of Gastroenterology, Aalborg Hospital, Aalborg, Denmark
- Department of Suregery, Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Bouwense SA, Olesen SS, Drewes AM, Poley JW, van Goor H, Wilder-Smith OH. Effects of pregabalin on central sensitization in patients with chronic pancreatitis in a randomized, controlled trial. PLoS One. 2012;7(8):e42096. doi: 10.1371/journal.pone.0042096. Epub 2012 Aug 6. PMID 22879908
- [Derived] Olesen SS, Graversen C, Olesen AE, Frokjaer JB, Wilder-Smith O, van Goor H, Valeriani M, Drewes AM. Randomised clinical trial: pregabalin attenuates experimental visceral pain through sub-cortical mechanisms in patients with painful chronic pancreatitis. Aliment Pharmacol Ther. 2011 Oct;34(8):878-87. doi: 10.1111/j.1365-2036.2011.04802.x. Epub 2011 Aug 16. PMID 21848870